CLINICAL TRIAL: NCT04874935
Title: The Possible Efficacy and Safety of Lansoprazole Co-administration With Neoadjuvant Chemotherapy in Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Samah Hussein Mohamed, Principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34615/4/21
Record Dates: First submitted 2021-04-29; First posted 2021-05-06 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lansoprazole arm (Active Comparator): 33 patients who will receive neoadjuvant chemotherapy and lansoprazole 60 mg twice daily four days before starting chemotherapy regimen and then the same dose will be used during chemotherapy cycles
  Interventions: Drug: Lansoprazole
- Placebo arm (Placebo Comparator): 33 patients who will receive neoadjuvant chemotherapy and placebo capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lansoprazole — administration of lansoprazole 60 mg twice daily 4 days before starting neoadjuvant chemotherapy regimen and continue till end of chemotherapy cycles
  Arms: Lansoprazole arm
Drug: Placebo — administration of Placebo capsule twice daily 4 days before starting neoadjuvant chemotherapy regimen and continue till end of chemotherapy cycles
  Arms: Placebo arm

SUMMARY:
Investigation of the possible efficacy and safety of lansoprazole co-administration with neoadjuvant chemotherapy in tumor response in women with breast cancer who will be planned for surgery.

DETAILED DESCRIPTION:
Several studies revealed that PPIs inhibit not only the H+/K+ ATPase in gastric parietal cells, but also the vacuolar H+ ATPase (V-ATPase) overexpressed in tumor cells, the V-ATPase is an ATP-dependent proton pump that transports H+ across both intracellular and plasma membranes to regulate intracellular and extracellular pH.

Co-administration or pretreatment with PPIs could inhibit H+ transport via the V-ATPase in tumor cells, resulting in lower extracellular acidification and intracellular acidic vesicles which increase the sensitivity of the tumor cells to the anticancer agents. Moreover, the low extracellular pH induces an increased activity of drug efflux pumps P-glycoprotein (P-gp), which is closely associated with multi-drug resistance (MDR) of tumors. As a consequence, there remains a lower concentration of chemotherapeutic drugs in tumor cells and reduced cytotoxic efficacy, thus restoring the normal extracellular PH will decrease MDR.

ELIGIBILITY:
Inclusion Criteria:

* Females with age ≥ 18 years old.
* Newly diagnosed breast cancer patients.
* Planned neoadjuvant chemotherapy.

Exclusion Criteria:

* Pregnancy.
* Nursing mothers.
* Active or uncontrolled infection.
* Presence of another malignancies.
* Inadequate blood picture.
* Serum Creatinine more than 1.5 mg /dl.
* AST and ALT more than 2.5 upper limit.
* History of known hypersensitivity to lansoprazole.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Tumor Response | 6 months
  - Tumor response evaluation will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Change in ki67 level | baseline and end of neoadjuvant chemotherapy cycles each cycle will be repeated every 21 days or may postponed according to patient condition and doctor instructions.
  - Assessment of the level of Ki-67 expression in cancer cells through a staining process (a marker of cancer cell proliferation).
Change in P-gp level | baseline and end of neoadjuvant chemotherapy cycles each cycle will be repeated every 21 days or may postponed according to patient condition and doctor instructions.
  - Assessment of P-gp level by ELISA Kits according to manufacturer's instructions.

SECONDARY OUTCOMES:
Adverse events and toxicity | 6 months
  - Adverse events and toxicity will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
Follow up of kidney function | baseline and monthly through study completion, an average of 4 to 6 months
  measurement of serum creatinine levels in (mg/dl) and blood urea nitrogen (BUN) levels in (mg/dl) from blood samples will be assessed monthly for all participants.
Follow up of liver function | baseline and monthly through study completion, an average of 4 to 6 months
  measurement of alanine transaminase (ALT) and aspartate transaminase (AST) both in U/L from blood samples will be assessed monthly for all participants.
Follow up of complete blood count | baseline and monthly through study completion, an average of 4 to 6 months
  measurement of the counts of red blood cells, white blood cells, platelets, hemoglobin and hematocrit will be assessed monthly for all participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Tanta, Egypt

REFERENCES:
- [Background] Lee YY, Jeon HK, Hong JE, Cho YJ, Ryu JY, Choi JJ, Lee SH, Yoon G, Kim WY, Do IG, Kim MK, Kim TJ, Choi CH, Lee JW, Bae DS, Kim BG. Proton pump inhibitors enhance the effects of cytotoxic agents in chemoresistant epithelial ovarian carcinoma. Oncotarget. 2015 Oct 27;6(33):35040-50. doi: 10.18632/oncotarget.5319. PMID 26418900
- [Background] Whitton B, Okamoto H, Packham G, Crabb SJ. Vacuolar ATPase as a potential therapeutic target and mediator of treatment resistance in cancer. Cancer Med. 2018 Aug;7(8):3800-3811. doi: 10.1002/cam4.1594. Epub 2018 Jun 21. PMID 29926527
- [Background] Ikemura K, Hiramatsu S, Okuda M. Drug Repositioning of Proton Pump Inhibitors for Enhanced Efficacy and Safety of Cancer Chemotherapy. Front Pharmacol. 2017 Dec 12;8:911. doi: 10.3389/fphar.2017.00911. eCollection 2017. PMID 29311921
- [Background] Lu ZN, Tian B, Guo XL. Repositioning of proton pump inhibitors in cancer therapy. Cancer Chemother Pharmacol. 2017 Nov;80(5):925-937. doi: 10.1007/s00280-017-3426-2. Epub 2017 Aug 31. PMID 28861639
- [Background] Wang BY, Zhang J, Wang JL, Sun S, Wang ZH, Wang LP, Zhang QL, Lv FF, Cao EY, Shao ZM, Fais S, Hu XC. Intermittent high dose proton pump inhibitor enhances the antitumor effects of chemotherapy in metastatic breast cancer. J Exp Clin Cancer Res. 2015 Aug 22;34(1):85. doi: 10.1186/s13046-015-0194-x. PMID 26297142
- [Background] da Silva VP, Mesquita CB, Nunes JS, de Bem Prunes B, Rados PV, Visioli F. Effects of extracellular acidity on resistance to chemotherapy treatment: a systematic review. Med Oncol. 2018 Oct 30;35(12):161. doi: 10.1007/s12032-018-1214-4. PMID 30377828